CLINICAL TRIAL: NCT07172308
Title: High Risk Atherosclerosis Identified at Cardiac CT Among Patients With vs Without Family History of CAD
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Elena Cittera, Head Scientific Direction, I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Other Study IDs: FRATER Study
Record Dates: First submitted 2025-08-31; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease (CAD); Atherosclerosis of Coronary Artery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute coronary syndrome often represtent the first drammatic manifestation of coronary atherosclerosis.

Cardiac computed tomography angiography (CCTA) has recently gained a pivotal role in the evalution of patients with suspected coronary artery disease (CAD). Of inteterst, it may provide important information on coronary atherosclerosis beyond lumen stenosis; more precisely high risk plaque features could be identified even in the abesence of significative lumen stenosis (i.e. not flow-limiting lesions).

The evidence of non-obstructive but high risk atheroscleorisis may support aggressive primary prevention treatment, reducing the risk of future cardiovascular events. Even if familty history of CAD is considered a risk factor for cardiovascular events, no clear data are available regarding the prevalence of coronary atherosclerosis in this subgroup of patients and CCTA in asymptomatic subjects is not clearly supported by evidence nor suggested by guidelines.

Aim of our study is to explore whether the prevalence of high risk coronary atherosclerosis among patients with family hystory of CAD is different when compared with a group of patients without family hystory of CAD.

For that purpose from consecutive registry of patient who underwent clinically indicated CCTA for suspected but unknown CAD a cohort of patients with family history of CAD as first early presentation of coronary atherosclerosis (group 1) will be compared with a consecutive cohort of subjects without familiy history of CAD (group 2). All CCTA will be perfomed according to most recent guidelines and advanced atheroscleoris analysis will be performed. As primary objective of the study, the prevalence of high risk atherosclerosis will be compared between the two Groups.

The evidence of higher prevalence of high-risk atherosclerosis prevalence in group 1 vs group 2 may further support the use of CCTA in asymptomatic patients but with family history of CAD.

ELIGIBILITY:
Inclusion Criteria:

* Group 1
* Patients with clinical indation to CCTA for suspected CAD with family history of CAD
* Age >40 years old for male and >50 years old for female
* No history of previous cardiovascular disease Group 2
* Patients with clinical indation to CCTA for suspected CAD without family history of CAD
* Age >40 years old for male and >50 years old for female
* No history of previous cardiovascular disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: History of any adverse reaction to contrast medium
  * History of any severe allergic reactions
  * Previous history of chronic kidney disease (eGFR<30 ml/min/1.73m2)
  * Previous history of cardiovascular disease, including documented asymptomatic atherosclerosis
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Identification of high risk atherosclerosis at coronary computed tomography angiography (CCTA) | Day 1
  the present is a trasveral descriptive study. No follow-up will be performed and all parameters will be evaluated at the time of CCTA acquisition (Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy

IPD SHARING:
Plan to Share IPD: No